CLINICAL TRIAL: NCT03502980
Title: Safety and Efficacy of Midline and Peripherally Inserted Central Catheter for Intravenous Therapy: a Randomized Controlled Trial
Brief Title: Safety and Efficacy of Midline and PICC
Acronym: MidLine_PICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7749
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2021-08

CONDITIONS: Vascular Access Devices; Central Venous Catheter
Keywords: Peripherally Inserted Central Catheter Line Insertion; Catheterization, Peripheral Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripherally inserted central venous catheters (Active Comparator): Bard PowerPICC
  Interventions: Device: Bard PowerPICC
- Midline (Active Comparator): Bard PowerMidline catheter
  Interventions: Device: Bard PowerMidline catheter

INTERVENTIONS:
Device: Bard PowerPICC — PICC Insertion
  Arms: Peripherally inserted central venous catheters
Device: Bard PowerMidline catheter — Midline Insertion
  Arms: Midline

SUMMARY:
The purpose of this study is to assess the non-inferiority for safety and efficacy of using Midline in comparison with PICC for intravenous therapy that do not require a central catheter.

DETAILED DESCRIPTION:
Vascular access devices (VADs), including peripherally inserted central venous catheters (PICCs) remain a cornerstone for the delivery of necessary intravenous therapy. PICCs are being selected for venous access more frequently today than ever before.

The advantage of PICC is that it can be used for all intravenous therapy. However, PICC requires the use of fluoroscopy or other type of guidance which add to the cost and time required to insert the catheter. Midline, on the other hand, can be inserted under ultrasound guidance, takes less time to be inserted and cost less than PICC insertion.

Despite lower cost and better accessibility of midline in comparison with PICC for non-vesicant intravenous therapy, there is very little evidence in the literature to suggest that one type of venous access is better than the other.

The primary objective of this study is to assess the non-inferiority for safety and efficacy of using Midline in comparison with PICC for intravenous therapy that do not require a central catheter.

Results of this trial will allow improving a quality of evidence for using midline instead of PICC for specified indications. If Midline are non-inferior for some indications, they would represent a more accessible and less expensive alternative than PICC insertion.

ELIGIBILITY:
Inclusion Criteria:

* Required intra venous therapy
* Expected duration of the venous access: > 6 days and < 30days

Exclusion Criteria:

* Patient has a contraindication to insertion of either a Midline or a PICC relative to the therapy
* Patient from other hospitals who come to the CHUM only for the installation of a central line
* Decreased cognitive ability to care for device at home
* Preexisting bacteremia (ie, existing positive blood cultures that had not been repeated with negative results)
* Preexisting venous thrombosis or known hypercoagulable states (such as protein C or S deficiency, antithrombin deficiency, lupus anticoagulant)
* Venous access with multiple lumens required
* Patients not able to give informed consent
* Prior participation to this study
* Patient is enrolled in another investigational study
* Patients hospitalized in the intensive care unit
* Patients who are difficult to puncture and require multiple blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
% of patients without VAD-related adverse event requiring medical intervention | Until 1 week after VAD retrieval
  Infections, Thrombophlebitis, Infiltration, Bleeding, Pain, Death
% of patients whose intended or additional I.V treatments could be completed with the VAD without VAD complications, dysfunctions or limitations (ex: need for central access or for additional peripheral or central lumens/catheters) | Until 1 week after VAD retrieval

SECONDARY OUTCOMES:
% of patients who experience VAD-related adverse events requiring medical intervention | Until 1 week after VAD retrieval
  Infections, Thrombophlebitis, Infiltration, Bleeding, Pain, Death
Number of VAD-related adverse events requiring medical intervention per 1000 catheter/days | Until 1 week after VAD retrieval
Time to first VAD-related adverse events | Until 1 week after VAD retrieval
Duration VAD intervention (Midline or PICC) | Index procedure
Number of additional interventions to insert the VAD | Index procedure
% of patients who required another VAD to complete the intended or additional iv treatments, either because of VAD complications, dysfunctions or limitations | Until 1 week after VAD retrieval
% of patient without failed blood sampling attempts through the VAD | Until 1 week after VAD retrieval
% of patients for whom the end of treatment was the reason for VAD retrieval | Until 1 week after VAD retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Éric Thérasse, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bentridi A, Giroux MF, Soulez G, Bouchard L, Perreault P, Chouinard A, Dorais M, Do Amaral R, Bernier P, Therasse E. Midline Venous Catheter vs Peripherally Inserted Central Catheter for Intravenous Therapy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e251258. doi: 10.1001/jamanetworkopen.2025.1258. PMID 40111366